CLINICAL TRIAL: NCT00213356
Title: Evoked Responses of External Anal Sphincter After Cortical and Lombo-sacral Magnetic Stimulations
Brief Title: Study of the Nervous Control of the Anal Sphincter
Status: Withdrawn | Type: Observational
Why Stopped: patients with neurological disease not included
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2001/099/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injuries - anal sphincter - evoked potentials
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anal incontinence and constipation are frequently observed in patients with neurological disease. The purpose of this study is to evaluate the neurological control of the anal sphincter in healthy subjects, patients with neurological disease by a new electrophysiological technique. This technique consists in recordings of anal sphincter responses after magnetic stimulations of the cortex and the sacral nerves.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* patients with spinal lesion
* patients with cauda equina syndrome

Exclusion Criteria:

* pregnant women
* pacemaker or other metallic material implanted
* epileptic patients
* organic colorectal disease
* obese patients
* previous neurological surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers patients with spinal lesion patients with cauda equina syndrome
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-04; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie LEROI, PHD, Principal Investigator — University Hospital, Rouen
Locations (1):
- University hospital of Rouen, Rouen, France